CLINICAL TRIAL: NCT00659087
Title: A Pilot Study of the Feasibility of Early Discharge After Total Knee Arthroplasty Using a Femoral Nerve Block
Brief Title: Effectiveness of a Femoral Block Following Total Knee Arthroplasty (TKA)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Edmonton Civic Employees Research Fund (Other)
Responsible Party: Principal Investigator, Tsui, Ban / Johnston DWC, Pediatric and Adult Anesthesiologist, Associate Professor/Director of Clinical Research, Stollery Children's Hospital/University of Alberta Hospital, Edmonton Civic Employees Research Fund
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: J-3224
Record Dates: First submitted 2008-04-10; First posted 2008-04-16 (Estimated); Last update posted 2016-08-03 (Estimated); Status verified 2016-08

CONDITIONS: Total Knee Arthroplasty
Keywords: Total Knee; Range of Motion; Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Femoral Block (Experimental): Those receiving femoral block in addition to usual pain management
  Interventions: Procedure: Femoral Block
- Usual Care (Active Comparator): Those receiving only usual pain management without a femoral block
  Interventions: Other: Usual Care

INTERVENTIONS:
Procedure: Femoral Block — Those receiving femoral block postoperatively
  Arms: Femoral Block
Other: Usual Care — Those receiving only usual pain management postoperatively
  Arms: Usual Care

SUMMARY:
Hospital stays after total joint replacement surgery have been getting shorter over the past 10 years. This is mostly due to new ways to manage pain and early rehabilitation. To be able to go home safely soon after surgery, patients need to:

* 1) have adequate pain control
* 2) be able to move through activities of daily living on their own (using aids)

Femoral nerve block, in combination with pain medications, is one of the new treatment strategies that are currently being used at other hospitals in Canada, the United States and the United Kingdom. Nerve blocks involve a needle filled with local anesthetic into the nerve that allows the feeling of pain around the knee. With good pain management, patients will be able to more quickly bend their knee and regain the ability to walk with aids and move from sitting and lying positions to standing and walking. Once they can do these activities with adequate pain control, they can be discharged from hospital to continue recovery at home. The purpose of this study is to examine a new way of managing postoperative pain and encourage early knee flexion and mobility, while maintaining pain control for patients after total knee replacement. We believe that patients who receive the nerve block in addition to the regular pain medication will have more knee flexion at discharge and experience less pain than patients who only receive usual pain medications.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing primary total knee arthroplasty
* English-speaking
* Preoperative knee ROM > 90 degrees
* Body Mass Index < 40

Exclusion Criteria:

* Regular preoperative opioid use
* Hepatic insufficiency
* Any contra-indications to receiving a femoral block

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-04; Primary Completion 2009-10 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
knee flexion | at hospital discharge or day 4 postoperatively, whichever is earlier

SECONDARY OUTCOMES:
pain | daily in hospital, 2 weeks, 6 weeks, 12 weeks
length of hospital stay | during hospitalization
nausea/vomiting | during hospitalization
participation in rehabilitation | day of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alberta Hospitals, Edmonton, Alberta, Canada